CLINICAL TRIAL: NCT00466388
Title: An Investigator-Initiated,Multicenter,Randomized,Double-Blind Placebo-Controlled Design Study to Assess the Effectiveness of CeviMeline to Improve OraL Health in Patients With XErostomia Secondary to Radiation Therapy for Treatment of Head and Neck Squamous Cell Carcinoma
Brief Title: Study of the Effectiveness of Cevimeline on Oral Health in Patients With Radiation Induced Xerostomia
Acronym: SMILE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Academy of Otolaryngology-Head and Neck Surgery Foundation (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAO-101
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Xerostomia
Keywords: dry mouth
MeSH Terms: conditions — Xerostomia | interventions — cevimeline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cevimeline (Experimental): Evoxac tid for xerostomia
  Interventions: Drug: Cevimeline
- Placebo (Placebo Comparator): sugar pill
  Interventions: Drug: Cevimeline

INTERVENTIONS:
Drug: Cevimeline
  Other Names: evoxac

SUMMARY:
The purpose of this study is to determine the effectiveness of cevimeline (versus placebo) on the oral health of patients who have dry mouth which was caused by radiation therapy that was given for treatment of head and/or neck cancer.

DETAILED DESCRIPTION:
Treatment of advanced head and neck squamous cell carcinoma (SCCA) requires aggressive therapy often combining surgical interventions with radiation therapy. Besides surveillance for persistent or recurrent cancer, clinicians seek to help minimize the side effects resulting from these aggressive treatments. Xerostomia, or "dry mouth", impacts each patient's long term health and quality of life due to the significant and diverse health consequences of having too little saliva. Normal swallowing, speaking, resistance to infection, and taste acuity are health domains that are affected by dry mouth. Psycho-social functioning decreases for many of these patients due to the extra effort to communicate and socialize (Locker D 2004).

Xerostomia is often a consequence of radiation treatment (XRT), especially when the XRT fields encompass the parotid glands and submandibular glands bilaterally. The disability and consequences of xerostomia extend beyond dysphagia, poor appetite secondary to difficulty of mastication, and loss of taste (Chambers et al. Xerostomia 2004). Since saliva is essential to normal oral flora and healthy teeth, the lack of saliva in these patients can dramatically and rapidly result in a decline of the patient's oral health. Dental complications can occur and present significant ongoing medical and surgical problems.

Our study proposes to use the Oral Health Impact Profile, OHIP-49, to measure disease-specific quality of life and functional outcomes due to radiation related xerostomia in head and neck cancer patients. The evaluation of patient QOL concomitantly with patient functioning as proposed in the SMILE protocol is an "evidence study to evaluate treatment effectiveness". The use of patient-oriented outcome measures are increasingly important to health insurers and government, but these measures are also aligned with the World Health Organization's mandate that health is a resource to manage which must be utilized and preserved so that individuals experience and gain satisfaction from living (Epstein J.1986). The OHIP-49 is patient reported outcome measure which is publicly available, validated in adult populations world-wide, and can be used an effectiveness measure. The questions are easy to answer and are based upon a 5 level likert type scale reflecting frequency of "bother" within individual psychosocial domains.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years old and able to give written informed consent
* Subject has received external beam radiotherapy > 4000 cGy for SCCA of the head and/or neck
* Radiation therapy was completed at least 16 weeks (4 months) prior to enrollment into the study but not greater than 52 weeks (12 months)
* Radiation included at least three of four of the major salivary glands (submandibular and parotid glands) in the initial field (boost fields may or may not include the parotid gland)
* Primary therapy was designed with curative intent. Surgery is permitted if the remaining inclusion criteria are met
* Grade 1 or 2 xerostomia by CTC version 3.0 criteria (Appendix D)
* Demonstratable salivary flow as assessed by the clinician after administration of a potent sialogogue such as lemon juice (1 teaspoon)
* Subject has at least one anatomically intact parotid gland and one submandibular gland
* ECOG performance status of 0, 1, or 2
* An EKG obtained has been performed in the past 6 months showing no arrhythmias or contraindication to administration of a muscarinic agent AND there has been no interval change in cardiac health
* Subject is able to eat an oral diet to maintain adequate hydration and nutrition
* Subject has provided informed consent
* Subject is English speaking and of sufficient mental capacity to comply with the study requirements
* Female subjects of child bearing potential have a negative serum pregnancy test and agree to use an approved method of birth control

Exclusion Criteria:

* Subject has a life expectancy less than 12 months.
* Subject is known or suspected to have persistent disease after curative intent
* Subject is greater than 12 months out from completion of radiation therapy
* Subject is pregnant or nursing
* Subject had previous cancer of the head and/or neck and is being treated with a second course of radiation therapy
* Subject has a history of an autoimmune disease with pretreatment xerostomia (i.e. Sjogrens) or other underlying systemic illness known to cause xerostomia independent of prior radiation therapy exposure
* Subject has had resection of both parotid glands
* Subject has history of cardiomyopathy or untreated moderate to severe CAD
* Subject has known cardiac arrhythmias
* Subject has grade 3 xerostomia (CTC v.3)or no demonstratable salivary flow after the test dose by visual inspection
* Subject has history of significant renal or hepatic impairment
* Subject uses a gastrostomy tube for nutrition supplementation
* Subject is taking medications specified in Appendix C
* Subject is taking or has taken any investigational new drug within the last 30 days or is planning to take such a drug during the course of this study
* Subject has a contraindication to administration of muscarinic medications.
* Subject has been treated previously with a muscarinic agent for xerostomia (i.e., Pilocarpine HCl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To assess the impact of increased salivary flow due to treatment with cevimeline compared to placebo in patient reported oral health using the OHIP-49 | 6 weeks

SECONDARY OUTCOMES:
To evaluate if increased salivary flow due to cevimeline treatment results in improved patient reported quality of life using the UW-QOL-HN | 6 weeks
To evaluate which subscales of the OHIP-49 are improved most by increased salivary flow due to cevimeline treatment | 6 weeks
To evaluate which subscales of the UW-QOL-HN are improved most by increased salivary flow due to cevimeline treatment | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Witsell, MD, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - Colorado Springs, Colorado
  - Carle Clinic Association, Urbana, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Commonwealth Ear, Nose and Throat, Louisville, Kentucky
  - Associated Otolaryngologist, Palmyra, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Fauquier ENT Consultants, Warrenton, Virginia